CLINICAL TRIAL: NCT05339607
Title: Endoscopic Resection of Papillary Adenomas; a Novel Treatment Algorithm to Prevent Recurrence - a Pilot-study (ERASE-pilot)
Acronym: ERASE-pilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Rogier P. Voermans, R.P. Voermans MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021.0684; NL79410.029.21 (Other: CCMO)
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Papillary Adenoma
Keywords: Endoscopic papillectomy; Recurrence; STSC; Intraductal ablation; Cystotome
MeSH Terms: conditions — Adenoma; Recurrence

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Other: Thermal ablation of resection margins by STSC and biliary orifice by cystotome.

INTERVENTIONS:
Other: Thermal ablation of resection margins by STSC and biliary orifice by cystotome. — Patients who are eligible will undergo thermal ablation of the resection margins.

SUMMARY:
Recurrence after endoscopic papillectomy is described in up to 33% of the cases (range 12-33%). This leads to re-interventions, a cumulative risk of adverse events, and the need for long-term follow-up. Recurrences most likely originate from either the biliary orifice or lateral resection margins. Ablative methods such as radiofrequency ablation (RFA) and thermal ablation by cystotome inside the bile duct have been described to treat intraductal extension of which the use of a cystotome seems to have a more favorable safety profile. However, no studies focusing on the preventive use of these ablative methods in patient with papillary adenomas have been performed. It is hypothesized that the curative resection rate can be increased and recurrence prevented by using a combination of snare tip soft coagulation (STSC) of the resection margins and thermal ablation by cystotome of the biliary orifice in patients with and without the suggestion of intraductal extension.

Therefore, aim of this study is to assess the safety and feasibility of endoscopic papillectomy combined with thermal ablation of the biliary orifice by cystotome and STSC of the lateral resection margins.

ELIGIBILITY:
Inclusion Criteria:

* Papillary adenoma which seems suitable for curative endoscopic resection.
* 18 years or older.
* Capable of providing written and oral informed consent.

Exclusion Criteria:

* Patients with intraductal extension of >1 cm beyond the duodenal wall or adenocarcinoma will be excluded since surgical resection is considered the preferred treatment in these cases.
* Failure to place a PD stent in patients with normal pancreatic duct anatomy.
* Refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety (rate of adverse events) | During 9 months follow-up
  i.e. pancreatitis, bleeding, cholangitis, perforation, and papillary stenosis.

SECONDARY OUTCOMES:
Curative resection rate | 3 and 9 months
  Defined as absence of adenomatous residual tissue or recurrence observed in follow-up biopsy sampling.
Additional yield of EUS prior to resection. | Prior to intervention.
  Intraductal growth or invasive growth encountered by EUS and not other imaging
Effect of hemospray as first modality in case of post procedural bleeding in need of intervention. | Delayed bleeding is expected not more than 30 days after the procedure
  Succesfull treatment of post procedural bleeding e.g. no need for re-intervention or transfusion.
Individual components of the primary outcome. | During 9 months follow-up
  i.e. rate of adverse events such as pancreatitis, bleeding, cholangitis, perforation, and papillary stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Rogier P Voermans, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No